CLINICAL TRIAL: NCT00938041
Title: Retreatment Study of Patients With Non-Hodgkin's Lymphoma Who Have Previously Responded to Iodine-131 Anti B1 Antibody
Brief Title: Retreatment of Patients With Non-Hodgkin's Lymphoma Who Have Previously Responded to Iodine-131 Anti B1 Antibody
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 393229/010
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

ARMS (1):
- Retreatment of NHL with Iodine-131 Anti-B1 Antibody (Experimental): Patients with non-Hodgkin's lymphoma who previously responded with a duration of response of at least 3 months to Iodine-131 Anti-B1 Antibody therapy will undergo two phases of study. In the first phase, patients will receive a dosimetric dose of unlabeled Anti-B1 Antibody (450 mg) followed by Anti-B1 Antibody (35 mg) which has been radiolabeled with 5 mCi of Iodine-131. Whole body gamma camera scans will be obtained after the dosimetric dose and data from three imaging time points will be used to calculate a patient-specific dose to deliver the desired total body dose of radiotherapy. In the second phase, patients will receive the therapeutic dose of unlabeled Anti-B1 Antibody (450 mg) followed by 35 mg of Anti-B1 Antibody labeled with the patient-specific dose to deliver the desired whole body dose of radiation. Patients will be treated with thyroid blocking medication at least 24 hours prior to the first infusion and continuing for 14 days following the last infusion.
  Interventions: Biological: Tositumomab and Iodine I 131 Tositumomab

INTERVENTIONS:
Biological: Tositumomab and Iodine I 131 Tositumomab — Tositumomab and Iodine I 131 Tositumomab

SUMMARY:
This multicenter study will determine the response rate, the complete response rate, duration of response, time to progression, time-to-treatment failure, safety, and survival following treatment with Iodine-131 Anti-B1 Antibody for the retreatment of patients with non-Hodgkin's lymphoma who previously responded with a duration of response of at least 3 months to Iodine-131 Anti-B1 Antibody therapy. Patients will undergo two phases of study. In the first phase, patients will receive a dosimetric dose of unlabeled Anti-B1 Antibody (450 mg) followed by Anti-B1 Antibody (35 mg) which has been radiolabeled with 5 mCi of Iodine-131. Whole body gamma camera scans will be obtained after the dosimetric dose and data from three imaging time points will be used to calculate a patient-specific dose to deliver the desired total body dose of radiotherapy. In the second phase, patients will receive the therapeutic dose of unlabeled Anti-B1 Antibody (450 mg) followed by 35 mg of Anti-B1 Antibody labeled with the patient-specific dose to deliver the desired whole body dose of radiation. Patients will be treated with thyroid blocking medication at least 24 hours prior to the first infusion and continuing for 14 days following the last infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed initial diagnosis of non-Hodgkin's B-cell lymphoma
* Patients must have previously responded with a duration of response of at least 3 months to Iodine-131 Anti-B1 Antibody therapy
* Patients must have evidence that their tumor tissue had CD20 expression
* Patients must have performance status of at least 60% on the Karnofsky scale and an anticipated survival of at least 3 months
* Patients must have absolute granulocyte count (ANC) greater than 1,500 cells/mm3 and platelet count greater than 100,000 cells/mm3 within 14 days of study entry without support of hematopoietic cytokines or transfusion of blood products
* Patients must have adequate renal (serum creatine less than 1.5 x upper limit of normal) and hepatic function (total bilirubin less than 1.5 x upper limit of normal and hepatic transaminases, AST and ALT, less than 5 x upper limit of normal) within 14 days of study entry
* Patients must have bi-dimensionally measurable disease with a least one lesion greater than or equal to 2 cm x 2 cm by CT scan
* Patients must be at least 18 years of age
* Patients must give written informed consent and sign an Institutional Review Board/Ethics Committee- approved informed consent form prior to study entry

Exclusion Criteria:

* Patients with more than 25% bone marrow involvement
* Patients who have received cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within 4 weeks prior to study entry or who exhibit persistent clinical evidence of toxicity. The use of systemic steroids much be discontinued at least 1 week prior to study entry.
* Patients with active obstructive hydronephoresis
* Patients with evidence of active infection requiring IV antibiotics at time of study entry
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease free for 5 years
* Patients with known HIV infection
* Patients with known brain or leptomeningeal metasteses
* Patients who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 1998-04; Primary Completion 2003-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 393229/010 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab: Participants were treated with a saturated solution of potassium iodide (KI), Lugol's solution, or KI tablets orally starting at least 24 hours prior to the first infusion of Iodine I-131 Tositumomab (TST) and continuing for 14 days following the last infusion of Iodine I-131 TST. Participants received treatment in two phases. The dosimetric dose was administered in Phase 1 as 450 milligrams (mg) of TST infused over 1 hour, followed by 35 mg of antibody containing 5 millicurie (mCi) of Iodine I-131 TST infused over 20 minutes (min), followed by a 10-min normal saline flush. The therapeutic dose, administered 7-14 days after the dosimetric dose, was administered as 450 mg of TST infused over 1 hour, followed by 35 mg of antibody radiolabeled with enough Iodine I-131 TST to deliver 75 centigrey (cGy) infused over 20 min, followed by a 10-min normal saline flush.
Period: Overall Study
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Started | 32
Completed | 5
Not Completed | 27
Not completed — Lost to Follow-up | 6
Not completed — Received Alternative Therapy | 1
Not completed — Progressive Disease | 5
Not completed — Death | 12
Not completed — Adrenal Insufficiency | 3

BASELINE CHARACTERISTICS:
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (12.5)
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response and Confirmed Complete Response
Description: Complete response (CR) is defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease. Response is defined as the best response achieved at any evaluation. A confirmed response is defined as a response that was confirmed by two separate response evaluations occurring at least 4 weeks apart.
Time Frame: Every 6 months until disease progression, death, or for 2 years following the dosimetric dose, whichever occurred first (average of 80.2 months)
Population: ITT-Exposed Population: all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 32
Participants
  Complete response | 8
  Confirmed complete response | 8
Statistical Analysis 1: Comparison: Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab; Test type: Superiority or Other; percentage of participants = 25, 95% CI 2-sided [10 to 40] — The estimated value reflects the percentage of participants with complete response. Percentages are calculated using the number of participants in the ITT-Exposed Population as the denominator
Statistical Analysis 2: Comparison: Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab; Test type: Superiority or Other; percentage of participants = 25, 95% CI 2-sided [10 to 40] — The estimated value reflects the percentage of participants with confirmed complete response. Percentages are calculated using the number of participants in the ITT-Exposed Population as the denominator

2. Primary Outcome: Duration of Response for All Confirmed Responders (CR + CCR + PR)
Description: For participants with CR, clinical CR (CCR), or partial response (PR), duration of response is defined as the time from the first documented response to the first documented progression. CCR is defined as the complete resolution of all disease-related symptoms, but residual foci, thought to be residual scar tissue, are present. Generally, an unchanging lesion <=2 centimeters (cm) in diameter by radiographic evaluation or <=1 cm in diameter by physical examination can be considered scar tissue. The extent of disease must be unchanged or decreased upon follow-up evaluations and, if unchanged or if further decreases for 6 months or longer are present, the participant will then be reclassified as a CR (complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease). PR is defined as a >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions, with no new lesions.
Time Frame: as for outcome 1
Population: ITT-Exposed Population. Only those participants with a confirmed CR, CCR, or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 18
Months | 18.9 [10.4 to 94.3]

3. Primary Outcome: Progression-free Survival
Description: Progression-free survival (time to progression or death) is defined as the time from the start of retreatment (i.e., the dosimetric dose) to the first documented progression or death. Disease Progression (PD) is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measurable lesions or the appearance of any new lesion. Individual lesions must be grater than 2 cm diameter by radiographic evaluation or grater than 1 cm diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT-Exposed Population. Participants who did not progress or die were censored at their date of last contact in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 32
Months | 11.9 [6.3 to 26.5]

4. Primary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from the dosimetric dose to the first occurrence of treatment withdrawal, a decision to receive additional therapy, study withdrawal, disease progression, or death.
Time Frame: as for outcome 1
Population: ITT-Exposed Population. Participants who withdrew from the study for reasons other than progression or death were censored at the date of study withdrawal. Participants who did not meet any of the criteria for treatment failure were censored at their date of last contact in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 32
Months | 11.7 [6.0 to 21.4]

5. Primary Outcome: Overall Survival
Description: Time to death (overall survival) is defined as the time from the start of retreatment (i.e., the dosimetric dose) to the date of death from any cause.
Time Frame: as for outcome 1
Population: ITT-Exposed Population. Participants who did not die were censored at the date of their last contact in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 32
Months | 64.2 [52.5 to 159.0]

6. Primary Outcome: Number of Participants With Any Serious Adverse Event (SAE) and Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as those events that were fatal or immediately life-threatening, and those events that resulted in hospitalization; prolonged an existing hospitalization; or resulted in disability, congenital anomaly, or cancer. Refer to the general AE/SAE module for a complete list of all AEs and SAEs.
Time Frame: as for outcome 1
Population: ITT-Exposed Population
Measure: Number; unit: Participants
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Number analyzed (Participants) | 32
Participants
  Any Adverse Event | 32
  Any Serious Adverse Event | 18

ADVERSE EVENTS:
Arm/Group | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab
Serious Adverse Events (participants affected / at risk) | 18/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab (N=32)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Caecitis (Gastrointestinal disorders) | 1
Lobar pneumonia (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Lymphomatoid papulosis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tositumomab and Antibody Radiolabeled Iodine I-131 Tositumomab (N=32)
Fatigue (General disorders) | 15
Asthenia (General disorders) | 6
Chills (General disorders) | 4
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 3
Pain (General disorders) | 2
Axillary pain (General disorders) | 1
Chest discomfort (General disorders) | 1
Local swelling (General disorders) | 1
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Tongue eruption (Gastrointestinal disorders) | 1
White blood cell < 2000 cells/mm^3 (Investigations) | 14
Absolute neutrophil count < 1000 cells/mm^3 (Investigations) | 12
Platelets < 50000 cells/mm^3 (Investigations) | 12
Hemoglobin < 8.0 grams/deciliter (Investigations) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Oral herpes (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Headache (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Mental impairment (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Axillary mass (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Lymphoedema (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Breath sounds abnormal (Investigations) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Diplopia (Eye disorders) | 1
Pupillary reflex impaired (Eye disorders) | 1
Strabismus (Eye disorders) | 1
Dysuria (Renal and urinary disorders) | 2
Stress urinary incontinence (Renal and urinary disorders) | 1
Tachycardia (Cardiac disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.